CLINICAL TRIAL: NCT02799147
Title: Dose-escalation Study of Graft-versus-host Disease Prophylaxis With High-dose Post-transplantation Bendamustine in Patients With Refractory Acute Leukemia
Brief Title: GVHD Prophylaxis With Post-transplantation Bendamustine in Refractory Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/16-n
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Leukemia, Acute Lymphoblastic; Acute Myeloid Leukemia; Mixed-Lineage Acute Leukemias
Keywords: Allogeneic Transplantation; Hematopoietic Stem Cell Transplantation; Leukemia, Acute Lymphoblastic; Acute Myeloid Leukemia; Mixed-Lineage Acute Leukemias; Immune System Diseases; Immunosuppressive Agents; Myeloablative Agonists; Busulfan; Fludarabine; Antineoplastic Agents, Alkylating; Bendamustine Hydrochloride
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Immune System Diseases | interventions — fludarabine phosphate; Busulfan; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 280 mg/m2 bendamustine (Experimental): 10 patients Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -6 through -3: Busulfan 1 mg/kg po qid №14 Day 0: Infusion of unmanipulated graft Day +3 and +4: Bendamustine 140 mg/m2/day iv.
  Interventions: Procedure: Allogeneic stem cell transplantation; Drug: Fludarabine monophosphate; Drug: Busulfan; Drug: Bendamustine
- 200 mg/m2 bendamustine (Experimental): 10 patients Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -6 through -3: Busulfan 1 mg/kg po qid №14 Day 0: Infusion of unmanipulated graft Day +3 and +4: Bendamustine 100 mg/m2/day iv
  Interventions: Procedure: Allogeneic stem cell transplantation; Drug: Fludarabine monophosphate; Drug: Busulfan; Drug: Bendamustine
- 140 mg/m2 bendamustine (Experimental): 10 patients Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -6 through -3: Busulfan 1 mg/kg po qid №14 Day 0: Infusion of unmanipulated graft Day +3, +4: Bendamustine 70 mg/m2/day iv.
  Interventions: Procedure: Allogeneic stem cell transplantation; Drug: Fludarabine monophosphate; Drug: Busulfan; Drug: Bendamustine

INTERVENTIONS:
Procedure: Allogeneic stem cell transplantation
  Other Names: HSCT
Drug: Fludarabine monophosphate
Drug: Busulfan
Drug: Bendamustine

SUMMARY:
Several groups have demonstrated very low incidence of acute and chronic graft-versus-host disease (GVHD) with post-transplantation cyclophosphamide (PTCy) in haploidentical, unrelated and related allogeneic stem cell transplantation (SCT). Nonetheless for majority of the grafts, except for 10/10 HLA-matched bone marrow, with this type of prophylaxis require concomitant administration of calcineurin inhibitors±MMF, which delays immune reconstitution and development of graft-versus-leukemia (GVL) effect. So, despite reduction of transplant-related mortality, use of PTCy doesn't lead to the reduction of relapse incidence. This is particularly important for relapsed or refractory acute leukemia patients, where, despite all efforts to intensify conditioning regimens, relapses after SCT occur in more than 50% of patients, and long-term survival rarely exceeds 10-20%. In preclinical model of haploidentical SCT the substitution of post-transplantation cyclophosphamide with bendamustine, led to comparable GVHD control, but significantly augmented GVL effect. To test this hypothesis and improve the outcome of allogeneic SCT in refractory acute leukemia patients we initiated a pilot trial with high-dose post-transplantation bendamustine for GVHD prophylaxis. The selection of doses is based on the previous dose-escalation studies. Additional immunosuppression could be added for mismatched grafts.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis: Acute Myeloblastic Leukemia Acute Lymphoblastic Leukemia Mixed-Lineage Acute Leukemias

* Disease, refractory to at list one course of induction chemotherapy or immunotherapy
* More than 5% clonal blasts in the bone marrow or peripheral blood at the time of inclusion
* Signed informed consent
* Matched related, 8-10/10 HLA-matched unrelated or haploidentical donor available. The HLA typing is performed by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* No second tumors
* No severe concurrent illness
* No previous autologous or allogeneic stem cell transplantations

Exclusion Criteria:

* Karnofsky index <70%
* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >1.5 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment, defined by CRP level >70 mg/L or positive procalcitonin in patient with adequate empirical antibacterial and antifungal therapy.
* Requirement for vasopressor support at the time of enrollment
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Engraftment rate | 60 days
  Engraftment is defined as the first of 3 consecutive days with an ANC>500 per μl and WBC>1000 per μl. Platelet engraftment is not mandatory for the endpoint.

SECONDARY OUTCOMES:
Relapse rate analysis | 365 days
Non-relapse mortality analysis | 365 days
Incidence of acute GVHD, grades II-IV | 180 days
Incidence of chronic GVHD, moderate and severe (NIH criteria) | 365 days
Overall survival analysis | 365 days
Event-free survival analysis | 365 days
Toxicity (NCI CTCAE 4.03) | 100 days
  Toxicity parameters based on NCI CTCAE 4.03 grades: hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), mucositis (attending physician assessment), hemorrhagic cystitis (attending physician assessment), cardiotoxicity (ECG, echocardiography). Additional toxicity parameters: incidence and severity of veno-occlusive disease, incidence of transplant-associated microangiopathy
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Boris V. Afanasyev, Professor, Study Director — St. Petersburg State Pavlov Medical University
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Consultations are ongoing about how IPD initiative fits the local law "About personal data 152-fz".

REFERENCES:
- [Background] Stokes J, Hoffman EA, Zeng Y, Larmonier N, Katsanis E. Post-transplant bendamustine reduces GvHD while preserving GvL in experimental haploidentical bone marrow transplantation. Br J Haematol. 2016 Jul;174(1):102-16. doi: 10.1111/bjh.14034. Epub 2016 Mar 31. PMID 27030315